CLINICAL TRIAL: NCT02565537
Title: A Prospective Randomized Comparison of the AMO CustomVue to the Alcon Wavelight in Patients Undergoing LASIK
Brief Title: High Resolution Wavefront-guided vs. Wavefront Optimized LASIK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Edward E. Manche, Principal Investigator, Stanford University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 34288
Record Dates: First submitted 2015-09-28; First posted 2015-10-01 (Estimated); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Nearsightedness; Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- iDesign WFG LASIK (Active Comparator): Wavefront-guided LASIK
  Interventions: Procedure: LASIK
- Wavelight WFO LASIK (Active Comparator): Wavefront-optimized LASIK
  Interventions: Procedure: LASIK

INTERVENTIONS:
Procedure: LASIK — WFG vs. WFO LASIK

SUMMARY:
The investigators are comparing outcomes of LASIK surgery using a high definition wavefront-guided laser to a wavefront-optimized laser in patients with nearsightedness with and without astigmatism.

DETAILED DESCRIPTION:
The patients will have a comprehensive eye examination once they express an interest in the study. This includes a slit lamp examination of the front of the eye and a dilated fundoscopic examination of the back of the eye. If there is any pathology noted that would exclude the patient from the study, then the investigators will inform the patient and make an appropriate referral. if the patient is deemed appropriate for the study after a comprehensive examination included computerized videokeratography, then they can be enrolled. The patient will undergo bilateral simultaneous eye surgery. Which eye is treated with the CustomVue and which eye is treated with Wavelight will be randomized so there is a 50% chance for either eye to receive one treatment. The patients will be seen on the day of surgery, post op day one, one month, three months, six months and one year. The patient will receive topical antibiotics in each eye for one week following the procedure. The patient will receive pred forte 1% ophthalmic drops for one week after treatment. The patient will also receive vigamox ophthalmic drops for four days after treatment. All of this is within the usual and customary standard of care for the treatment of patients undergoing LASIK surgery.

ELIGIBILITY:
Inclusion criteria.

* Subjects age 21 and older with healthy eyes.
* Nearsightedness between -0.25 diopters and -11.00 diopters with or without astigmatism of up to 5.00 diopters.

Exclusion criteria.

* Subjects under the age of 21.
* Patients with excessively thin corneas.
* Patients with topographic evidence of keratoconus.
* Patients with ectatic eye disorders.
* Patients with autoimmune diseases.
* Patients who are pregnant or nursing.
* Patients must have similar levels of nearsightedness and farsightedness in each eye. They can not be more than 1.5 diopter of difference between eyes.
* Patients must have similar levels of astigmatism in each eye. They can not have more than 1.5 diopter of difference between eyes.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Uncorrected visual acuity | Twelve months

SECONDARY OUTCOMES:
Quality of vision and quality of life using the QoV questionnaire | One month, three months, six months and twelve months
Changes in higher order aberrations (Coma, trefoil, spherical aberration, total higher order RMS) | One day, one month, three months, six months and twelve months
Predictability of refractive outcomes (Percentage of eyes +/- 0.25 diopters, +/- 0.50 diopters and +/- 1.00 diopters of the intended correction) | One, three, six and twelve months
Change in best spectacle corrected visual acuity | One, three, six and twelve months
Vector analysis of astigmatic outcomes (The Alpins method looking at Target induced astigmatism, Surgical induced astigmatism, Index of Success | One, three six and twelve months

CONTACTS AND LOCATIONS:
Overall Officials: Edward E. Manche, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States

REFERENCES:
- [Background] Chiang B, Valerio GS, Manche EE. Prospective, Randomized Contralateral Eye Comparison of Wavefront-Guided Laser In Situ Keratomileusis and Small Incision Lenticule Extraction Refractive Surgeries. Am J Ophthalmol. 2022 May;237:211-220. doi: 10.1016/j.ajo.2021.11.013. Epub 2021 Nov 14. PMID 34788593